CLINICAL TRIAL: NCT07334158
Title: Effect of Critical Thinking Disposition Program on Developing Reflective Thinking and Motivation to Learn Among Nursing Students
Acronym: CTDP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MU-FN-CTDP-2026
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Critical Thinking; Reflective; Motivation; Nursing Students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention Group (Experimental): This group consists of nursing students who will participate in the Critical Thinking Disposition Program. The study included a single-arm group of 243 nursing students enrolled in the1st and 2nd year at [Technical Institute of Nursing / Mansoura University]. All participants were selected based on inclusion criteria of no prior exposure to critical thinking programs and willingness to participate
  Interventions: Other: Critical thinking disposition program

INTERVENTIONS:
Other: Critical thinking disposition program — structured educational intervention designed to enhance reflective thinking skills and motivation to learn. The program includes multiple interactive sessions focusing on critical analysis, problem-solving, decision-making, and self-reflection activities. Students will engage in exercises that encourage them to evaluate clinical scenarios, reflect on their learning experiences, and apply critical thinking strategies in practical nursing situations. The aim is to measure the program's impact on students' reflective thinking ability, critical thinking disposition, and learning motivation compared to their baseline levels. All participants will follow the standard nursing curriculum in addition to the intervention

SUMMARY:
Study Title:

Effect of Critical Thinking Disposition Program on Developing Reflective Thinking and Motivation to Learn among Nursing Students

Study Description:

This study aims to investigate the effect of a Critical Thinking Disposition Program on nursing students' reflective thinking and motivation to learn. In the rapidly evolving healthcare environment, nurses must possess both critical thinking skills and disposition to make accurate clinical judgments and provide high-quality professional care. Many novice nurses lack critical thinking disposition, which can result in inaccurate clinical judgments and an inability to identify causes of problems.

The program will target nursing students to enhance their internal motivation to think critically, solve problems, evaluate ideas, and make informed decisions. The intervention focuses on developing cognitive strategies, attitudes, and behaviors that support self-motivated learning and professional competence. Outcomes will be measured by evaluating students' reflective thinking and motivation to learn before and after the program.

Primary Outcome Measures:

Improvement in reflective thinking scores

Increase in motivation to learn scores

Secondary Outcome Measures:

Development of critical thinking disposition attributes such as truth-seeking, open-mindedness, analyticity, inquisitiveness, self-confidence, and maturity

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate and able to attend all program sessions.

No prior exposure to critical thinking training programs.

Exclusion Criteria:

* Students with learning difficulties or any limitations that prevent active participation in the program.

Students who miss more than 50% of the program sessions.

Students participating in external programs aimed at enhancing critical thinking during the study period.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 243 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reflective thinking | Before and 2 months after critical thinking disposition program
  Improvement in reflective thinking among nursing students, measured using the [name of validated questionnaire], assessed before and after the interventi

SECONDARY OUTCOMES:
Motivation to Learn | measured at baseline (pre-intervention) and immediately after completion of the program (post-intervention)
  Enhancement in students' learning motivation, evaluated using a validated motivation-to-learn scale

IPD SHARING:
Plan to Share IPD: Undecided